CLINICAL TRIAL: NCT04426955
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Camrelizumab (SHR-1210) Versus Placebo in Combination With Concurrent Chemoradiotherapy in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Study of Camrelizumab (SHR-1210) in Combination With Concurrent Chemoradiotherapy in Locally Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-323
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Cancer
Keywords: PD-1Antibody; locally advanced esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Paclitaxel; Cisplatin; Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Camrelizumb + Paclitaxel + Cisplatin + Radiotherapy.
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiation
- Arm B (Placebo Comparator): Placebo + Paclitaxel + Cisplatin + Radiotherapy.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Placebo; Radiation: Radiation

INTERVENTIONS:
Drug: Camrelizumab — IV infusion
  Other Names: SHR-1210
  Arms: Arm A
Drug: Paclitaxel — IV infusion
Drug: Cisplatin — IV infusion
Drug: Placebo — IV infusion
  Arms: Arm B
Radiation: Radiation — Concurrent Radiation

SUMMARY:
This is a randomised, double-blinded, placebo-controlled, multi-center phase III trial, comparing the efficacy and safety of treatment with Camrelizumab (SHR-1210) + definitive chemoradiotherapy(dCRT) vs placebo+dCRT for locally advanced esophageal cancer patients in China. Camrelizumab (SHR-1210) is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subjects will be randomized into study arm or control arm. Participants receive camrelizumab or placebo + chemotherapy + radiation therapy . The chemotherapy regimens are : paclitaxel plus cisplatin Progression-free survival (PFS) assessed by the Independent Review Committee (IRC) will be the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years; 2.Histologically confirmed diagnosis of localized ESCC; 3.Measurable and/or non-measurable disease defined per RECIST v1.1; 4.ECOG Performance Status ≤ 1; 5.Adequate organ function

Exclusion Criteria:

1. Indicators of severe malnutrition;
2. A history of surgery for esophageal cancer;
3. Clinically uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention;
4. Known to be intolerable or resistant to treatment with the protocol-specified chemotherapy;
5. Received prior chemotherapy, radiotherapy, targeted therapy or immune-oncology therapies;
6. Active autoimmune diseases or history of autoimmune diseases that may relapse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRC | up to 3 years
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
PFS assessed by investigators | up to 3 years
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
OS | up to 3 years
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive. Measured by the method of Kaplan and Meier.
ORR | up to 3 years
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
DoR | up to 3 years
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
AE | up to 3 years
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No